CLINICAL TRIAL: NCT05824182
Title: Fostering Resilience and Well-being in Young Adults With a History of Adverse Childhood Experiences - the FACE Self-help App
Brief Title: The FACE Self-help App for Fostering Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeannette Brodbeck (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor-Investigator, Jeannette Brodbeck, Prof. Dr., University of Applied Sciences and Arts Northwestern Switzerland
Organization: University of Applied Sciences and Arts Northwestern Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SNF_197731_B
Record Dates: First submitted 2023-03-23; First posted 2023-04-21 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Adverse Childhood Experiences
Keywords: Adverse Childhood Experiences; Psychosocial Functioning; Emotion Regulation; Social Information Processing; Online self-help
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention group: FACE self-help app with guidance
  Interventions: Device: FACE self-help App
- control group (No Intervention): Waiting list control group with questionnaires and EMA

INTERVENTIONS:
Device: FACE self-help App — The FACE self-help app was developed based on well-established non-invasive psychological principles that have been used in other web-based self-help interventions. The app consists of two component, emotion regulation and social information processing/social skills with four modules each. Each module includes readings describing scientific knowledge about ACEs and ACEs related topics, as well as exercises to encourage participants to actively reflect on what was learned in the readings and to apply their knowledge and practice skills. Each module is divided in several submodules that include readings and exercises.
  Arms: Intervention Group

SUMMARY:
The FACE self-help app is an online intervention for young adults with Adverse Childhood Experiences (ACEs). It was developed based on well-established cognitive-behavioural therapy principles. The self-help app contains two components, one targeting emotion regulation (ER), the other social information processing (SIP).

DETAILED DESCRIPTION:
The FACE self-help app is an online intervention for young adults with Adverse Childhood Experiences (ACEs). It was developed based on well-established cognitive-behavioural therapy principles. The self-help app contains two components, one targeting emotion regulation (ER), the other social information processing (SIP).

The goal of the present study is to evaluate the efficacy of the FACE self-help app, which aims to foster resilience and improve well-being by enhancing emotion regulation, social skills and minimizing biases in social information processing.

The primary objective is to examine the efficacy of the FACE self-help app for improving resilience and well-being in young adults with a history of ACEs compared to a waiting list control group and to examine the stability of a possible effect.

Secondary objectives are to test

1. the differential efficacy of the self- and emotion regulation and the social skills and social information processing component
2. the effects of the FACE self-help app on real life data in affective states, social interactions, the use of coping strategies and state resilience.

To assess real life data, additionally to questionnaires (Q), an ecological momentary assessment (EMA) will be conducted in three one-week episodes, with 6 daily assessments each.

Procedures: After giving informed consent, participants will receive the online questionnaires and one week of EMA (t0, week 1). Then, participants will be randomly assigned to either the intervention or waiting list control group. Within the intervention group, participants are randomly assigned to start with the ER or SIP component. After 5 weeks of using the first component of the FACE self-help app, participants fill out the intermediate measure (t1, week 7). After another week of EMA, the next component (ER or SIP) of the self-help app is available for 5 weeks. Subsequently, the post-measurement and the last EMA period start (t2, week 13). This results in a total intervention period of 11 weeks. A follow-up measure will be conducted after another 11 weeks (t4, week 25). Participants will receive online guidance from trained e-coaches.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported ACEs
* An informed consent
* The possession of a smartphone
* Mastery of the German language.
* Age between 18 and 25

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g., due to comprehension problems, visual impairment, lack of sufficient motor skills or severe psychological or somatic disorders which require immediate treatment which impedes the continuous work on the self-help programme. These points will be discussed with the participant in the screening telephone call.
* Acute suicidality.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 167 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Resilience | at week 13, t2 (post-measurement)
  Resilience will be assessed with the German version (Sarubin et al., 2015) of the Connor-Davidson Resilience Scale (CD-RISC) (Connor & Davidson, 2003). The scale contains 10 items that are rated on a 5-point scale from 0 - Not true at all to 4 - True nearly all the time. A higher score indicates more resilience.

SECONDARY OUTCOMES:
Well-being | at week 13, t2 (post-measurement)
  Well-being will be assessed with the Warwick-Edinburgh Mental Well-being Scale (WEMWBS) (Tennant et al., 2007). The scale contains 14 items that are rated on a 5-point scale from 1 - never to 5 - always. A higher score indicates better well-being.
Emotion Regulation | at week 13, t2 (post-measurement)
  Self-Efficacy for Managing Emotions will be assessed with the PROMIS Short Form v1.0 - Self-Efficacy for Managing Emotions (PROMIS, 2022). The scale contains 7 items that are rated on a 5-point scale from 1 - never to 5 - always. A higher score indicates better emotion regulation skills.
Fear of Negative Evaluation | at week 13, t2 (post-measurement)
  Fear of Negative Evaluation will be assessed with the German short version of the fear of Negative Evaluation Scale (SANB-5) (Kemper et al., 2012). The scale contains 5 items that are rated on a 4-point likert scale from 1 - almost never true to 4- almost always true. A higher score indicates more fear of negative evaluation.
Social Avoidance | at week 13, t2 (post-measurement)
  Social avoidance will be assessed with the subscale social-behavioral avoidance from the German version of the cognitive-behavioral avoidance scale (KBVS) (Röthlin et al., 2010). The subscale contains 8 items that are rated on a 5-point likert scale from 1 - not at all applicable for me to 5 - absolutely applicable for me. A higher score indicates more social avoidance.
Problem-Solving | at week 13, t2 (post-measurement)
  Problem-solving will be assessed with German version (Graf, 2003) of the short form of the Social Problem-Solving Inventory-Revised (SPSI-R) (D'Zurilla et al., 2002).The scale contains 25 items that are rated on a 5-point scale from 0 - not at all true to 4 - extremely true. The scale contains 5 subscales: positive problem orientation, negative problem orientation, rational problem-solving, impulsive style, avoidance style. A higher score indicates a higher orientation on each subscale.
Self-Esteem | at week 13, t2 (post-measurement)
  Self-esteem will be assessed with the German version (Collani & Herzberg, 2003) of the Rosenberg Self-Esteem Scale (Rosenberg, 1965). The scale contains 10 items that are rated on a 4-point scale from 1 - not at all true to 4 - extremely true. A higher score indicates more self-esteem.
Stability of improvement in well-being | at week 24, t4 (follow-up)
  Well-being will be assessed with the Warwick-Edinburgh Mental Well-being Scale (WEMWBS) (Tennant et al., 2007). The scale contains 14 items that are rated on a 5-point scale from 1 - never to 4 - always. A higher score indicates better well-being.
Stability of improvement in emotion regulation | at week 24, t4 (follow-up)
  Self-Efficacy for Managing Emotions will be assessed with the PROMIS Short Form v1.0 - Self-Efficacy for Managing Emotions (PROMIS, 2022). The scale contains 7 items that are rated on a 5-point scale from 1 - never to 5 - always. A higher score indicates better emotion regulation skills.
Stability of decrease in fear of negative evaluation | at week 24, t4 (follow-up)
  Fear of Negative Evaluation will be assessed with the German short version of the fear of Negative Evaluation Scale (SANB-5) (Kemper et al., 2012). The scale contains 5 items that are rated on a 4-point likert scale from 1 - almost never true to 4- almost always true. A higher score indicates more fear of negative evaluation.
Stability of decrease in social avoidance | at week 24, t4 (follow-up)
  Social avoidance will be assessed with the subscale social-behavioral avoidance from the German version of the cognitive-behavioral avoidance scale (KBVS) (Röthlin et al., 2010). The subscale contains 8 items that are rated on a 5-point likert scale from 1 - not at all applicable for me to 5 - absolutely applicable for me. A higher score indicates more social avoidance.
Stability of improvement in problem-solving | at week 24, t4 (follow-up)
  Problem-solving will be assessed with German version (Graf, 2003) of the short form of the Social Problem-Solving Inventory-Revised (SPSI-R) (D'Zurilla et al., 2002). The scale contains 25 items that are rated on a 5-point scale from 0 - not at all true to 4 - extremely true. The scale contains 5 subscales: positive problem orientation, negative problem orientation, rational problem-solving, impulsive style, avoidance style. A higher score indicates a higher orientation on each subscale.
Stability of improvement in self-esteem | at week 24, t4 (follow-up)
  Self-esteem will be assessed with the German version (Collani & Herzberg, 2003) of the Rosenberg Self-Esteem Scale (Rosenberg, 1965). The scale contains 10 items that are rated on a 4-point scale from 1 - not at all true to 4 - extremely true. A higher score indicates more self-esteem.
Stability of improvement in resilience | at week 24, t4 (follow-up)
  Resilience will be assessed with the German version (Sarubin et al., 2015) of the Connor-Davidson Resilience Scale (CD-RISC) (Connor & Davidson, 2003). The scale contains 10 items that are rated on a 5-point scale from 0 - Not true at all to 4 - True nearly all the time. A higher score indicates more resilience.

OTHER OUTCOMES:
Participant satisfaction | at week 13, t2 (post-measurement)
  The ZUF-8 is a self-report measure that explores patients' overall satisfaction with the treatment (Schmidt et al., 1989). For this study, the instrument was adapted to explore patients' satisfaction with the Internet intervention studied in this trial. The scale contains eight items that are rated on a 4-point scale from 1 - low satisfaction to 4 - high satisfaction. A higher score indicates more satisfaction with the online intervention. The German version of the ZUF-8 showed adequate psychometric properties with good internal consistency, construct validity, and concurrent validity (Schmidt et al., 1989).
Momentary affect | three one week periods with 6 measurements a day (t0, t1, t2)
  The scale is an abbreviated version of the PANAS following previous research, that used similar EMA items (Oorschot et al., 2013; Wichers et al., 2012).
Momentary coping | three one week periods with 6 measurements a day (t0, t1, t2)
  The items of the coping scale were developed by this research team on the basis of previous research (Daros et al., 2019). They measure different emotion regulation and coping strategies such as reappraisal, avoidance or changing the situation.
Momentary burden | three one week periods with 6 measurements a day (t0, t1, t2)
  These items were developed by this research team as an addition to the emotion regulation items based on feedback from a user testing group. The participants indicate how burdened they feel in different areas.The scale contains 6 items (school/work, family, friends, feelings/thoughts, difficult memories, leisure time) that are rated on a 7-point scale from 0 - not at all to 6 - extremely. Furthermore, participants can indicate burdens in other areas.
Momentary social interactions | three one week periods with 6 measurements a day (t0, t1, t2)
  These items were developed by this research team. The Items explore the participants emotional state in the last social situation, for example how happy a person felt in the interaction.
  First, participants are asked, if they had a social interaction since the last measurement. If participants indicate an interaction, there are 7 follow-up questions about how the participant felt in this interaction. The scale contains 7 items (stressed, well, anxious, understood, irritated, insecure, happy) that are rated on a 7-point scale from 0 - not at all to 6 - extremely.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette Brodbeck, Professor, Principal Investigator — University of Applied Sciences and Arts Northwestern Switzerland
Locations (1):
- University of Applied Sciences and Arts Northwestern Switzerland, Olten, Canton of Solothurn, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available on request to interested researchers
Supporting Information: Study Protocol
Time Frame: After the end of data collection (2025)
Access Criteria: Access to these data is permitted for scientific purposes on request. A data access agreement will be signed and the source of the data (including the funding agency) needs to be acknowledged.

REFERENCES:
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Daros, A. R., Daniel, K. E., Meyer, M. J., Chow, P. I., Barnes, L. E., & Teachman, B. A. (2019). Impact of social anxiety and social context on college students' emotion regulation strategy use: An experience sampling study. Motivation and Emotion, 43(5), 844-855. https://doi.org/10.1007/s11031-019-09773-x
- [Background] D'Zurilla, T. J., Nezu, A. M., & Maydeu-Olivares, A. (2002). Social problem-solving inventory-revised: Technical manual. North Tonawanda, NY: Multi-Health Systems, 475.
- [Background] Graf, A. (2003). Psychometrische Überprüfung einer deutschsprachigen Übersetzung des SPSI-R. Zeitschrift für Differentielle und Diagnostische Psychologie, 24(4), 277-291. https://doi.org/10.1024/0170-1789.24.4.277
- [Background] Grosse Holtforth, M., & Grawe, K. (2003). Der Inkongruenzfragebogen (INK). Zeitschrift für Klinische Psychologie und Psychotherapie, 32(4), 315-323. https://doi.org/10.1026/0084-5345.32.4.315
- [Background] Oorschot M, Lataster T, Thewissen V, Lardinois M, Wichers M, van Os J, Delespaul P, Myin-Germeys I. Emotional experience in negative symptoms of schizophrenia--no evidence for a generalized hedonic deficit. Schizophr Bull. 2013 Jan;39(1):217-25. doi: 10.1093/schbul/sbr137. Epub 2011 Oct 20. PMID 22021660
- [Background] PROMIS. (2022). https://www.healthmeasures.net/explore-measurement-systems/promis
- [Background] Rosenberg, M. (1965). Society and the adolescent self-image. Princeton university press.
- [Background] Sarubin, N., Gutt, D., Giegling, I., Bühner, M., Hilbert, S., Krähenmann, O., Wolf, M., Jobst, A., Sabaß, L., Rujescu, D., Falkai, P., & Padberg, F. (2015). Erste Analyse der psychometrischen Eigenschaften und Struktur der deutschsprachigen 10- und 25-Item Version der Connor-Davidson Resilience Scale (CD-RISC). Zeitschrift für Gesundheitspsychologie, 23(3), 112-122. https://doi.org/10.1026/0943-8149/a000142
- [Background] Schick M, Schonbucher V, Landolt MA, Schnyder U, Xu W, Maier T, Mohler-Kuo M. Child Maltreatment and Migration: A Population-Based Study Among Immigrant and Native Adolescents in Switzerland. Child Maltreat. 2016 Feb;21(1):3-15. doi: 10.1177/1077559515617019. Epub 2015 Nov 19. PMID 26590238
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Vormbrock, F., & Neuser, J. (1983). Konstruktion zweier spezifischer Trait-Fragebogen zur Erfassung von Angst in sozialen Situationen (SANB und SVSS). Diagnostica, 29(2), 165-182.
- [Background] Watson D, Friend R. Measurement of social-evaluative anxiety. J Consult Clin Psychol. 1969 Aug;33(4):448-57. doi: 10.1037/h0027806. No abstract available. PMID 5810590
- [Background] Wichers M, Peeters F, Rutten BP, Jacobs N, Derom C, Thiery E, Delespaul P, van Os J. A time-lagged momentary assessment study on daily life physical activity and affect. Health Psychol. 2012 Mar;31(2):135-44. doi: 10.1037/a0025688. Epub 2011 Oct 10. PMID 21988094
- [Background] Kemper, C. J., Lutz, J., & Neuser, J. (2012). Konstruktion und Validierung einer Kurzform der Skala Angst vor negativer Bewertung (SANB-5). Klinische Diagnostik und Evaluation, 4, 343-360.
- [Background] Röthlin, P., Holtforth, M. G., Bergomi, C., Berking, M., Ottenbreit, N. D., & Caspar, F. (2010). Vermeidung und depression. Diagnostica.
- [Derived] Brodbeck J, Botschi SIR, Vetsch N, Stallmann L, Lochner J, Berger T, Schmidt SJ, Marmet S. Fostering resilience and well-being in emerging adults with adverse childhood experiences: study protocol for a randomized controlled trial to evaluate the FACE self-help app. BMC Psychol. 2024 Feb 19;12(1):84. doi: 10.1186/s40359-024-01560-9. PMID 38374126